CLINICAL TRIAL: NCT03379545
Title: Preoperative Magnetic Resonance as an Alternative to Computed Tomography Three-Dimensional Imaging for Characterizing Bone Loss in Shoulder Arthroplasty Candidates With Glenohumeral Osteoarthritis: A Prospective, Blinded, and Controlled Clinical Trial.
Brief Title: 3D MR Versus 3D CT for Glenohumeral Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17-00500
Record Dates: First submitted 2017-12-07; First posted 2017-12-20 (Actual); Results first posted 2020-04-16 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Arthritis; Glenohumeral Osteoarthritis
MeSH Terms: conditions — Arthritis | interventions — Magnetic Resonance Imaging; Diagnostic Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- 3D MR and 3D CT Imaging (Other): All shoulder arthroplasty candidates with glenohumeral osteoarthritis will be receiving both 3D computed tomography (CT) and 3D non-contrast magnetic resonance (MR) imaging.
  Interventions: Diagnostic Test: 3-dimensional (3D) magnetic resonance (MR) imaging; Diagnostic Test: 3D computed tomography (CT) imaging

INTERVENTIONS:
Diagnostic Test: 3-dimensional (3D) magnetic resonance (MR) imaging — MRI is performed using 3T scanners with a dedicated 16-channel shoulder array coils. The MRI sequences include 3-mm slice thickness and 0.5-mm gap width with a field of view of 14 or 15 cm. There were 6 diagnostic sequences with axial, coronal, and sagittal proton density weighting as well as coronal T2 with frequency selective fat suppression and sagittal T1 images.
Diagnostic Test: 3D computed tomography (CT) imaging — The CT protocol consists of 3-mm axial images of the glenoid reconstructed into 1-mm sagittal and coronal 2D reconstructions using the following parameters: 120 kV, 280 mA, and pitch of 0.9. The CT data were also used to produce a 3D reconstruction of each glenoid.

SUMMARY:
This study aims to assess the efficacy of three-dimensional magnetic resonance (MR) compared to three-dimensional computed tomography (CT) imaging. This proposed study is a prospective, unrandomized, single-blinded, self-controlled, and single-armed diagnostic radiological evaluation study.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from glenohumeral OA;
* Radiographic evidence of severe glenoid erosion;
* Indication for TSA based on clinical exam;
* Patient is willing to participate by complying with pre-operative visit requirements;
* Patient is willing and able to review and sign a study informed consent form.

Exclusion Criteria:

* Prior arthroplasty at the affected shoulder;
* Patients with inflammatory arthritis;
* Patients with post-capsulorrhaphy arthritis;
* Patients with post-traumatic arthritis;
* Patients with rotator cuff tear arthropathy;
* Patients exhibiting a lack of physical or mental ability to perform or comply with the study procedures;
* Patients who are pregnant;
* Patients with implanted medical devices that are contraindicated to exposure up to a 3.0-tesla magnetic field.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-01-11 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2020-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph D Zuckerman, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Shoulder Arthroplasty (SA): 3D computed tomography (CT) and 3D non-contrast magnetic resonance (MR)
  3-dimensional (3D) magnetic resonance (MR): MRI is performed using 3T scanners with a dedicated 16-channel shoulder array coils. The MRI sequences include 3-mm slice thickness and 0.5-mm gap width with a field of view of 14 or 15 cm. There were 6 diagnostic sequences with axial, coronal, and sagittal proton density weighting as well as coronal T2 with frequency selective fat suppression and sagittal T1 images.
  3D computed tomography (CT) imaging: The CT protocol consists of 3-mm axial images of the glenoid reconstructed into 1-mm sagittal and coronal 2D reconstructions using the following parameters: 120 kV, 280 mA, and pitch of 0.9. The CT data were also used to produce a 3D reconstruction of each glenoid.
Period: Overall Study
Arm/Group | Shoulder Arthroplasty (SA)
Started | 29
Completed | 29
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Shoulder Arthroplasty (SA)
Number analyzed (Participants) | 29
Age, Continuous [Median (Full Range); unit: years] | 68 [47 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Glenoid Version
Description: All scans from 3D CT and 3D MR imaging were reviewed carefully for the presence of any morphological changes. For the determination of glenoid version, a line was drawn between the anterior and posterior margins of the glenoid. The transverse axis of the scapula was determined by a line drawn from the midpoint of the genoid fossa to the medial end of the image of the scapula; a line drawn perpendicular to this was defined as a line of neutral version. The angle between the line of neutral version and the line connecting the anterior and posterior margins of the glenoid was measured and recorded as the Glenoid Version.
Time Frame: 3 Months
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Shoulder Arthroplasty (SA)
Number analyzed (Participants) | 29
degrees
  3D-MR Scan | 12.1 (8.7)
  3D-CT Scan | 11.4 (7.4)

2. Primary Outcome: Glenoid Inclination
Description: The 3D MRI glenoid inclination is measured by the two observers with the same method used for CT 3D glenoid inclination measurement following generating a new 2D axial MR images form the 3D MRI model using the three-point method. A line on the supraspinatus fossa and 3 points are drawn: Point S represents the inferior border of the glenoid, point R represents the intersection of the supraspinatus fossa line with the glenoid surface, and point A represents the vertex of the right triangle created by the line of the supraspinatus fossa and a perpendicular line passing through point S; this line (RS) is the hypotenuse of the right triangle. The inclination corresponds to the area in which the glenoid component of RSA is implanted.
Time Frame: 3 Months
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | 3D MR and 3D CT Imaging
Number analyzed (Participants) | 29
degrees
  3D-MR Scan | 89.2 (7.2)
  3D-CT Scan | 91 (8.1)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Shoulder Arthroplasty (SA)
All-Cause Mortality (participants affected / at risk) | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-11): https://cdn.clinicaltrials.gov/large-docs/45/NCT03379545/Prot_SAP_000.pdf